CLINICAL TRIAL: NCT04465396
Title: A Randomized, Open-label, Two-treatment, Two-period, Single-dose, Crossover Study to Evaluate the Bioavailability of Teduglutide Administered Subcutaneously by Syringe Injection Versus Pen Injector in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Bioavailability of Teduglutide Administered Subcutaneously by Syringe Injection Versus Pen Injector in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-633-1001
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — teduglutide; Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cohort 1 (Teduglutide 3 mg): Treatment A1, Then Treatment B1 (A1B1) (Experimental): Teduglutide, 3 mg, subcutaneous (SC) injection using a syringe, once on Day 1 of Treatment Period 1 (Treatment A1), followed by same dose SC pen injector, once on Day 1 of Treatment Period 2 (Treatment B1). A Washout Period of 7 days was maintained between Treatment Periods 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
  Interventions: Drug: Teduglutide; Device: Syringe Injection; Device: Pen injector
- Cohort 1 (Teduglutide 3 mg): Treatment B1, Then Treatment A1 (B1A1) (Experimental): Teduglutide, 3 mg, SC pen injector, once on Day 1 of Treatment Period 1 (Treatment B1), followed by same dose SC injection using a syringe, once on Day 1 of Treatment Period 2 (Treatment A1). A Washout Period of 7 days was maintained between the Treatment Periods 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
  Interventions: Drug: Teduglutide; Device: Syringe Injection; Device: Pen injector
- Cohort 2 (Teduglutide 4 mg): Treatment A2, Then Treatment B2 (A2B2) (Experimental): Teduglutide, 4 mg, SC injection using a syringe, once on Day 1 of Treatment Period 1 (Treatment A2), followed by same dose SC pen injector, once on Day 1 of Treatment Period 2 (Treatment B2). A Washout Period of 7 days was maintained between Treatment Periods 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
  Interventions: Drug: Teduglutide; Device: Syringe Injection; Device: Pen injector
- Cohort 2 (Teduglutide 4 mg): Treatment B2, Then Treatment A2 (B2A2) (Experimental): Teduglutide, 4 mg, SC pen injector, once on Day 1 of Treatment Period 1 (Treatment B2), followed by same dose SC injection using a syringe, once on Day 1 of Treatment Period 2 (Treatment A2). A Washout Period of 7 days was maintained between Treatment Periods 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
  Interventions: Drug: Teduglutide; Device: Syringe Injection; Device: Pen injector

INTERVENTIONS:
Drug: Teduglutide — Participants received 3 mg or 4 mg of Teduglutide SC syringe injection followed by pen injector or vice versa depending upon the treatment sequence AB or BA on Day 1 of Treatment Periods 1 and 2.
  Other Names: TAK-633
Device: Syringe Injection — Teduglutide was administered using syringe.
Device: Pen injector — Teduglutide was administered using pen injector.

SUMMARY:
The purpose of this study is to evaluate the bioavailability of teduglutide administered as a single subcutaneous (SC) fixed dose (depending upon participant weightband assignment) delivered by a syringe injection and the same fixed dose delivered by the pen injector in healthy participants.

DETAILED DESCRIPTION:
This is a 2-period crossover study and consists of two cohorts. Cohort 1 consists of participant's with greater than or equal to (>=) 40.0 kilogram (kg) to lesser than or equal to (<=) 75.0 kg of weight and Cohort 2 consists of participant's with greater than (>) 75.0 kg to <= 120.0 kg of weight. Participants in each cohort will be randomized to 1 of 2 treatment sequences AB or BA. Randomization will be stratified by injection site (i.e., thigh, abdomen, and arm) within each cohort.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated informed consent and assent as applicable to participate in the study.
* Aged 18 - 45 inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a full physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, coagulation (as appropriate), serum chemistry, and urinalysis.
* Body mass index (BMI) >= 18.0 and l<=32.0 kilogram per square meter (kg/m^2) at screening. Body weight for a participant in Cohort 1 will be >= 40.0 kg to <= 75.0 kg, and body weight for a participant in Cohort 2 will be > 75.0 kg to <= 120.0 kg, inclusive. This inclusion criterion will be assessed at the screening visit and confirmed at first check-in.

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Positive PCR (polymerase chain reaction) test for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), either with the absence or presence of the clinical symptoms of Coronavirus disease 2019 (COVID-19).
* Known or suspected intolerance or hypersensitivity to teduglutide, closely-related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of teduglutide.
* Known history of alcohol or other substance abuse within the last year prior to screening.
* Donation of blood or blood products (e.g. plasma or platelets) within 60 days prior to receiving the first dose of teduglutide.
* Pregnant or lactating female.
* Within 30 days prior to the first dose of teduglutide:

  1. Have used an investigational product (if elimination half-life is lesser than [<] 6 days, otherwise 5 half-lives)
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's (or designee's) opinion, may impact this study
  3. Have had any substantial changes in eating habits, as assessed by the investigator (or designee)
* Use of dipeptidyl peptidase 4 inhibitors within 30 days or 5 half-lives, whichever is greater, prior to administration of the first dose of teduglutide.
* Confirmed systolic blood pressure > 140 millimeter of mercury (mmHg) or < 90 mmHg, and diastolic blood pressure > 90 mmHg or < 40 mmHg at screening.
* Twelve-lead electrocardiogram (ECG) demonstrating QTcF > 450 milliseconds (msec) at screening. If the QTcF exceeds the aforementioned limits, the ECG should be repeated 2 more times and the average of the 3 QTcF values should be used to determine the participants eligibility.
* Positive screen for drugs of abuse or alcohol at screening and at each check-in.
* Male participants who consume more than 21 units of alcohol per week or regularly consume more than 3 units per day. Female participants who consume more than 14 units of alcohol per week or regularly consume more than 2 units per day. (1 alcohol unit=150 milliliter [mL] of wine, or 360 mL of beer, or 45 mL of 45 percent [%] alcohol).
* Positive Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen at screening.
* Use of tobacco in any form (e.g. smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch) based on participant self-reporting. Ex-users must report that they have stopped using tobacco for at least 3 months prior to receiving the first dose of teduglutide.
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches. One caffeine unit is contained in the following items: one 6 ounce (oz) (180 mL) cup of coffee, two 12 oz (360 mL) cans of cola, one 12 oz (360 mL) cup of tea, three 1 oz (85 gram [g]) chocolate bars.
* Prior screen failure, randomization, participation, or enrollment in this study, or prior exposure to any Glucagon-like peptide 2 (GLP-2) analogs.
* Presence of lesions, rashes, tattoos, and moles etc. on administration sites not allowing adequate conduct of injection site reaction and injection site injury assessment
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations; with the exception of occasional use of ibuprofen [1.2 g per 24 hour period] or acetaminophen [2 g per 24 hour period]). Current use is defined as use within 14 days of the first dose of teduglutide and throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b600d4db2bf003ab48ce5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 13 January 2021 to 20 August 2021.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 2 cohorts of this 2-period cross-over study to receive teduglutide (TAK-633) 3 or 4 milligrams (mg), subcutaneously by syringe injection (Treatment A1 for Cohort 1 and Treatment A2 for Cohort 2) or through pen injector (Treatment B1 for Cohort 1 and Treatment B2 for Cohort 2). Randomization was stratified by injection site (thigh, abdomen, and arm) within each cohort .
Period: Treatment Period 1 (Day 1)
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1, Then Treatment B1 (A1B1) | Cohort 1 (Teduglutide 3 mg): Treatment B1, Then Treatment A1 (B1A1) | Cohort 2 (Teduglutide 4 mg): Treatment A2, Then Treatment B2 (A2B2) | Cohort 2 (Teduglutide 4 mg): Treatment B2, Then Treatment A2 (B2A2)
Started | 16 | 16 | 16 | 16
Completed | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1, Then Treatment B1 (A1B1) | Cohort 1 (Teduglutide 3 mg): Treatment B1, Then Treatment A1 (B1A1) | Cohort 2 (Teduglutide 4 mg): Treatment A2, Then Treatment B2 (A2B2) | Cohort 2 (Teduglutide 4 mg): Treatment B2, Then Treatment A2 (B2A2)
Started | 16 | 16 | 16 | 16
Completed | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 1)
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1, Then Treatment B1 (A1B1) | Cohort 1 (Teduglutide 3 mg): Treatment B1, Then Treatment A1 (B1A1) | Cohort 2 (Teduglutide 4 mg): Treatment A2, Then Treatment B2 (A2B2) | Cohort 2 (Teduglutide 4 mg): Treatment B2, Then Treatment A2 (B2A2)
Started | 16 | 16 | 16 | 16
Completed | 16 | 15 | 15 | 16
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1, Then Treatment B1 (A1B1) | Cohort 1 (Teduglutide 3 mg): Treatment B1, Then Treatment A1 (B1A1) | Cohort 2 (Teduglutide 4 mg): Treatment A2, Then Treatment B2 (A2B2) | Cohort 2 (Teduglutide 4 mg): Treatment B2, Then Treatment A2 (B2A2) | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 64
Age, Continuous [Mean (Full Range); unit: years] | 31.8 [20 to 41] | 32.4 [20 to 45] | 32.5 [18 to 39] | 35.9 [23 to 45] | 33.2 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 2 | 1 | 21
  Male | 7 | 7 | 14 | 15 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 9 | 9 | 42
  Not Hispanic or Latino | 6 | 2 | 7 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 3 | 11
  White | 12 | 14 | 10 | 13 | 49
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 16 | 16 | 64
Height [Mean (Full Range); unit: cm] | 163.19 [151.0 to 175.0] | 164.06 [151.0 to 177.0] | 173.81 [165.0 to 189.0] | 175.38 [163.0 to 187.0] | 169.11 [151 to 189]
Weight [Mean (Full Range); unit: kg] | 64.38 [55.4 to 73.5] | 66.51 [55.8 to 73.4] | 86.39 [74.9 to 108.8] | 84.68 [75.3 to 106.8] | 75.49 [55.4 to 108.8]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2]
  kg/m^2 | 24.271 [19.31 to 30.72] | 24.891 [20.12 to 30.25] | 28.558 [23.98 to 31.81] | 27.530 [22.99 to 31.41] | 26.313 [19.31 to 31.81]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Verse Time Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-last) of Teduglutide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: Pharmacokinetic (PK) Set included all participants who received at least one dose of the study drug and have at least 1 quantifiable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Groups:
- Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection): Teduglutide, 3 mg, SC injection using a syringe, once on Day 1 of Treatment Period 1 and 2 (Treatment A1). Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector): Teduglutide, 3 mg, SC pen injector, once on Day 1 of Treatment Period 1 and 2 (Treatment B1). Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection): Teduglutide, 4 mg, SC injection using a syringe, once on Day 1 of Treatment Period 1 and 2 (Treatment A2). Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector): Teduglutide, 4 mg, SC pen injector, once on Day 1 of Treatment Period 1 and 2 (Treatment B2). Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng*hour/mL | 217.2 (21.0) | 237.2 (22.1) | 221.9 (21.2) | 253.0 (21.4)
Statistical Analysis 1: Comparison: Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) vs Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector); Test type: Equivalence — Equivalence between pen injector and syringe injection was to be considered established if the 90% confidence interval (CI) of the corresponding geometric mean ratio was within the acceptance interval of 80.00% to 125.00%; Geometric Mean Ratio = 109.22, 90% CI 2-sided [104.83 to 113.80] — The analysis was performed using Proc Mixed in statistical software suite (SAS), with treatment, sequence, period, and participant within sequence as fixed effects
Statistical Analysis 2: Comparison: Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) vs Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector); Test type: Equivalence — Equivalence between pen injector and syringe injection was to be considered established if the 90% CI of the corresponding geometric mean ratio was within the acceptance interval of 80.00% to 125.00%; Geometric Mean Ratio = 113.99, 90% CI 2-sided [108.32 to 119.95] — The analysis was performed using Proc Mixed in SAS, with treatment, sequence, period, and participant within sequence as fixed effects

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Teduglutide
Description: Cmax is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: PK Set included all participants who received at least one dose of the study drug and have at least 1 quantifiable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
ng/mL | 33.90 (37.7) | 33.31 (37.6) | 31.99 (34.8) | 29.58 (32.6)
Statistical Analysis 1: Comparison: Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) vs Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 98.27, 90% CI 2-sided [88.50 to 109.11] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) vs Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 92.48, 90% CI 2-sided [83.80 to 102.05] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) of Teduglutide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: PK Set included all participants who received at least one dose of the study drug and have at least 1 quantifiable plasma concentration. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 30 | 30 | 30 | 30
ng*hr/mL | 227.6 (21.1) | 249.2 (20.8) | 227.1 (20.8) | 268.2 (22.2)
Statistical Analysis 1: Comparison: Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) vs Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 109.44, 90% CI 2-sided [105.51 to 113.51] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) vs Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 118.40, 90% CI 2-sided [112.31 to 124.83] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Area Under the Plasma Concentration Verse Time Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-last) of Teduglutide by Injection Site
Description: AUC0-last of teduglutide by injection site (i.e., thigh, abdomen, and arm) was assessed and reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Cohort 1 (Teduglutide 3 mg): Syringe Injection in Abdomen: Teduglutide, 3 mg, SC injection using a syringe in the abdomen, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Syringe Injection in Arm: Teduglutide, 3 mg, SC injection using a syringe in the arm, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Syringe Injection in Thigh: Teduglutide, 3 mg, SC injection using a syringe in the thigh, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Pen Injector in Abdomen: Teduglutide, 3 mg, SC pen injector in the abdomen, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Pen Injector in Arm: Teduglutide, 3 mg, SC pen injector in the arm, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 1 (Teduglutide 3 mg): Pen Injector in Thigh: Teduglutide, 3 mg, SC pen injector in the thigh, once on Day 1 of Treatment Period 1 and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 2 (Teduglutide 4 mg): Syringe Injection in Abdomen: Teduglutide, 4 mg, SC injection using a syringe in the abdomen, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Syringe Injection in Arm: Teduglutide, 4 mg, SC injection using a syringe in the arm, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Syringe Injection in Thigh: Teduglutide, 4 mg, SC injection using a syringe in the thigh, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Pen Injector in Abdomen: Teduglutide, 4 mg, SC pen injector in the abdomen, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Pen Injector in Arm: Teduglutide, 4 mg, SC pen injector in the arm, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
- Cohort 2 (Teduglutide 4 mg): Pen Injector in Thigh: Teduglutide, 4 mg, SC pen injector in the thigh, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
Arm/Group | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Abdomen | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Arm | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Thigh | Cohort 1 (Teduglutide 3 mg): Pen Injector in Abdomen | Cohort 1 (Teduglutide 3 mg): Pen Injector in Arm | Cohort 1 (Teduglutide 3 mg): Pen Injector in Thigh | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Abdomen | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Arm | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Thigh | Cohort 2 (Teduglutide 4 mg): Pen Injector in Abdomen | Cohort 2 (Teduglutide 4 mg): Pen Injector in Arm | Cohort 2 (Teduglutide 4 mg): Pen Injector in Thigh
Number analyzed (Participants) | 12 | 10 | 10 | 12 | 10 | 10 | 12 | 10 | 10 | 12 | 10 | 10
ng*hr/mL | 241.2 (14.0) | 205.8 (29.1) | 202.2 (14.4) | 277.6 (9.1) | 216.6 (27.8) | 215.2 (16.7) | 219.6 (17.2) | 222.6 (27.9) | 224.1 (20.3) | 239.5 (19.0) | 277.3 (23.3) | 246.4 (21.3)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Teduglutide by Injection Site
Description: Cmax of teduglutide by injection site (i.e., thigh, abdomen, and arm) was assessed and reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Abdomen | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Arm | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Thigh | Cohort 1 (Teduglutide 3 mg): Pen Injector in Abdomen | Cohort 1 (Teduglutide 3 mg): Pen Injector in Arm | Cohort 1 (Teduglutide 3 mg): Pen Injector in Thigh | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Abdomen | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Arm | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Thigh | Cohort 2 (Teduglutide 4 mg): Pen Injector in Abdomen | Cohort 2 (Teduglutide 4 mg): Pen Injector in Arm | Cohort 2 (Teduglutide 4 mg): Pen Injector in Thigh
Number analyzed (Participants) | 12 | 10 | 10 | 12 | 10 | 10 | 12 | 10 | 10 | 12 | 10 | 10
ng/mL | 40.84 (29.7) | 31.66 (41.6) | 29.02 (35.2) | 43.65 (20.7) | 28.73 (43.9) | 27.91 (27.3) | 26.86 (25.9) | 38.28 (43.8) | 32.97 (25.0) | 28.14 (30.4) | 32.33 (33.8) | 28.73 (35.5)

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) of Teduglutide by Injection Site
Description: AUC0-infinity of teduglutide by injection site (i.e., thigh, abdomen, and arm) was assessed and reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Cohort 1 (Teduglutide 3 mg): Syringe Injection in Abdomen: Teduglutide, 3 mg, SC injection using a syringe in the abdomen, once on Day 1 of Treatment Period 1and 2. Participants with >=40.0 kg to <=75.0 kg of weight were included in Cohort 1.
- Cohort 2 (Teduglutide 4 mg): Syringe Injection in Thigh: Teduglutide, 4 mg, SC injection using a syringe in the thigh, once on Day 1 of Treatment Period 1 and 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.Teduglutide, 4 mg, SC injection using a syringe in the abdomen, once on Day 1 of either Treatment Period 1 or Treatment Period 2. Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
Arm/Group | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Abdomen | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Arm | Cohort 1 (Teduglutide 3 mg): Syringe Injection in Thigh | Cohort 1 (Teduglutide 3 mg): Pen Injector in Abdomen | Cohort 1 (Teduglutide 3 mg): Pen Injector in Arm | Cohort 1 (Teduglutide 3 mg): Pen Injector in Thigh | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Abdomen | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Arm | Cohort 2 (Teduglutide 4 mg): Syringe Injection in Thigh | Cohort 2 (Teduglutide 4 mg): Pen Injector in Abdomen | Cohort 2 (Teduglutide 4 mg): Pen Injector in Arm | Cohort 2 (Teduglutide 4 mg): Pen Injector in Thigh
Number analyzed (Participants) | 12 | 9 | 9 | 12 | 9 | 9 | 12 | 9 | 9 | 12 | 9 | 9
ng*hr/mL | 246.6 (13.2) | 213.0 (29.5) | 218.6 (18.7) | 282.3 (9.1) | 229.6 (26.8) | 229.2 (18.6) | 224.7 (17.6) | 228.2 (27.1) | 228.7 (20.0) | 247.0 (19.7) | 296.8 (24.4) | 268.1 (20.9)

7. Secondary Outcome: Time of First Occurrence of Maximum Observed Plasma Concentration (Cmax) [Tmax] of Teduglutide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
hour | 4.002 [2.00 to 8.06] | 4.001 [0.50 to 8.05] | 4.999 [2.01 to 8.04] | 4.507 [2.00 to 12.00]

8. Secondary Outcome: Terminal Disposition Phase Rate Constant (Lambda z) of Teduglutide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 30 | 30 | 30 | 30
1/hr | 0.4055 (51.2) | 0.4191 (41.0) | 0.3971 (41.8) | 0.3236 (48.1)

9. Secondary Outcome: Terminal Disposition Phase Half-Life (t1/2z) of Teduglutide
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 30 | 30 | 30 | 30
hour | 1.930 (1.1070) | 1.797 (0.8341) | 1.903 (0.9107) | 2.385 (1.2292)

10. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Teduglutide
Description: CL/F for extravascular administration divided by the fraction of dose absorbed of teduglutide was assessed and reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter(L)/hr
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 30 | 30 | 30 | 30
Liter(L)/hr | 13.48 (3.2060) | 12.31 (2.9332) | 17.97 (3.5737) | 15.27 (3.5042)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Teduglutide
Description: Vz/F associated with the terminal slope following extravascular administration divided by the fraction of dose absorbed of teduglutide was assessed and reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24 hours post-dose of Treatment Period 1 and Treatment Period 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 30 | 30 | 30 | 30
L | 36.85 (18.837) | 31.86 (15.382) | 49.84 (27.394) | 51.01 (23.867)

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an AE that started or worsened at the time of or after study drug administration. Number of participants with TEAEs included injection site reactions and injection site injury assessments.
Time Frame: From the start of study drug administration up to follow-up (up to 42 days)
Population: Safety Set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 13 | 10 | 9 | 5

13. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Vital signs included body temperature, respiratory rate, blood pressure, and heart rate.
Time Frame: From the start of study drug administration up to follow-up (up to 42 days)
Population: Safety Set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Clinical laboratory assessments included hematology, serum chemistry, coagulation, and urinalysis. Changes in laboratory values may be considered as AE if they were judged to be clinically significant.
Time Frame: From the start of study drug administration up to follow-up (up to 42 days)
Population: Safety Set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examination included examination of respiratory, cardiovascular, and gastrointestinal system.
Time Frame: From the start of study drug administration up to follow-up (up to 42 days)
Population: Safety Set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection)): Teduglutide, 4 mg, SC injection using a syringe, once on Day 1 of Treatment Period 1 and 2 (Treatment A2). Participants >75.0 kg to <=120.0 kg of weight were included in Cohort 2.
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection)) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Device Malfunction
Description: Number of participants with device malfunction was assessed and reported. The site staff reported any malfunctions whilst using the device.
Time Frame: Day 1
Population: Safety Set included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to follow-up (up to 42 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. AEs were collected and reported as per Treatment (A1, B1, A2, and B2) throughout the study.
Arm/Group | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 13/32 | 10/32 | 9/32 | 1/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Teduglutide 3 mg): Treatment A1 (Syringe Injection) (N=32) | Cohort 1 (Teduglutide 3 mg): Treatment B1 (Pen Injector) (N=32) | Cohort 2 (Teduglutide 4 mg): Treatment A2 (Syringe Injection) (N=32) | Cohort 2 (Teduglutide 4 mg): Treatment B2 (Pen Injector) (N=32)
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 1 | 2 | 0
Injection site pain (General disorders) | 2 | 1 | 3 | 1
Vessel puncture site pain (General disorders) | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04465396/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04465396/SAP_001.pdf